CLINICAL TRIAL: NCT00137072
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose Parallel Study of Men With Mild to Moderate Erectile Dysfunction to Evaluate the Efficacy of Viagra 8 Hours Post-Dose
Brief Title: Mild To Moderate Erectile Dysfunction Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481230
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Viagra (Sildenafil Citrate) 100 mg

SUMMARY:
Safety/Efficacy of 100-mg Viagra at 8 hours post dose in men with mild to moderate erectile dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Men 18-70 years of age
* Documented clinical diagnosis of erectile dysfunction of at least 3 months duration.

Exclusion Criteria:

* Subjects with penile implants
* Subjects with a known history of retinitis pigmentosa.
* Subjects, due to the requirement of 100 mg dosage, who are receiving concomitant treatment with the potent CYP3A4 inhibitor ritonavir.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2005-04; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of sexual intercourses that are successful in men with mild to moderate ED 8 hrs after a dose of Viagra.

SECONDARY OUTCOMES:
To determine the proportion of sexual intercourses that are successful in men with mild to moderate ED 12 hrs after a dose of Viagra. Other questionnaires such as SEP, IIEF.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Homewood, Alabama
  - Pfizer Investigational Site, Hoover, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Middlebury, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Hattiesburg, Mississippi
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Bay Shore, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Lacey, Washington
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481230&StudyName=Mild+To+Moderate+Erectile+Dysfunction+study